CLINICAL TRIAL: NCT05255068
Title: Optimizing Mealtime Care (OPTIMAL): Development and Pilot Testing of a Person-Centered Mealtime Care Intervention for Nursing Home Residents With Alzheimer's Disease and Related Dementias (ADRD)
Brief Title: OPTIMAL in NH Residents With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Wen Liu, Associate Professor, University of Iowa
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: K23AG066856 (NIH); K23AG066856 (NIH)
Record Dates: First submitted 2022-01-17; First posted 2022-02-24 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Alzheimer's Disease and Related Dementias
Keywords: Alzheimer's Disease and Related Dementias; Mealtime; Eating; Behavioral Symptoms; Food Intake; Function; Nutrition; Nursing Homes
MeSH Terms: conditions — Alzheimer Disease; Behavioral Symptoms | interventions — Optimal Pressed Ceramic

STUDY DESIGN:
Masking Description: Because this study is a single-group design, all participants were recruited from the nursing home site that was assigned as the intervention group. no one is blinded to the intervention assignment, but all participants and outcome assessors were blinded for the research questions/aims.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Staff (Experimental): Start participants who enrolled in the study, received the OPTIMAL intervention, and were observed during data collection.
  Interventions: Behavioral: OPTIMAL
- Resident (Experimental): Resident participants who were cared in the study site, and received care from the staff participants before and after the OPTIMAL intervention was delivered to staff.
  Interventions: Behavioral: OPTIMAL

INTERVENTIONS:
Behavioral: OPTIMAL — A person-centered mealtime care intervention

SUMMARY:
The purpose of this study is to develop and refine OPTIMAL and evaluate its feasibility, fidelity, and usefulness. The OPTIMAL is designed to teach staff to effectively engage residents in eating using individualized, person-centered behavioral strategies.

DETAILED DESCRIPTION:
This study developed and refined OPTIMAL, and evaluated its feasibility, fidelity, and usefulness. We used mixed methods (i.e., focus groups, a pilot single-group repeated measures) to refine and test OPTIMAL. We collected repeated measures at 3 time points: baseline (T1), immediately post intervention (6 weeks post baseline, T2), and 6-week post intervention (12 weeks post baseline, T3). At each time point, we assessed quality of staff engagement and resident outcomes including eating performance and BMI through collection and coding of videotaped observations of dyadic mealtime interaction (videos; Aim 2&3) over 6 meals in 2 consecutive days (2 breakfasts, 2 lunches, 2 dinners) for each staff-resident dyad. We used Cue Utilization and Engagement in Dementia (CUED) mealtime video coding scheme, an innovative, feasible, and reliable tool that our team has developed and validated, and assessed resident mealtime challenging behaviors including resistive behaviors and functional impairments and intake success rate using videos collected in this study.11, 25

The specific aims are:

1. Develop, evaluate, and refine OPTIMAL intervention protocol and training materials. We will integrate evidence from literature and our prior work to develop the intervention protocol and training materials, addressing resident mealtime difficulties, targeted PCMC strategies, and establishment of individualized PCMC plans. We will conduct separate focus group interviews of staff and family participants on the acceptability and appropriateness of the intervention protocol and training materials before pilot testing. Data obtained will be used to refine the intervention protocol and training materials before pilot testing.
2. Determine feasibility, fidelity, and usefulness of OPTIMAL. Feasibility on participant identification, recruitment, consent, and retention will be evaluated descriptively. Fidelity will be assessed on a) delivery of treatment (staff attendance to training sessions), b) receipt of treatment (staff knowledge and self-efficacy pre- & post-training), and c) enactment of treatment skills (staff PCMC&TCMC behaviors, quality of staff engagement). We will conduct focus group interviews of staff to assess the usefulness of OPTIMAL after T3.
3. Describe resident outcomes (Exploratory). We will measure and describe resident mealtime difficulties, eating performance, intake success rate, body weight, and body mass index using descriptive statistics over time for two treatment groups. Data obtained will inform estimates of effect sizes for a future larger-scale trial.

ELIGIBILITY:
The investigators will recruit direct care staff, families of residents, and residents with dementia from NH sites following the exclusion and inclusion criteria after attrition rates are considered.

Inclusion Criteria:

Residents

* ≥ 55 years
* Diagnosed as having ADRD based on medical records
* Identified by NH staff as requiring mealtime assistance
* Having a legally authorized representative (LAR) providing informed written consent

Staffs

* ≥18 years
* English speaking
* A permanent facility employee
* Provide direct mealtime care for a resident participant at least twice a week over the previous month

Families

* ≥18 years
* English speaking
* A family member of the resident who is living at the NH study site at the time of the study
* Having experience of delivering mealtime care to their resident family members

Exclusion Criteria:

Residents

* Have a documented diagnosis of Parkinson's disease, traumatic brain injury, or swallowing disorder,
* Do not eat orally (e.g., parenteral/IV feedings, feeding tubes)
* Unable to hear or see staff even with glasses and/or hearing aids (e.g., uncorrected visual or hearing impairment)
* Stay in the NH study site for less than 12 weeks at the time of recruitment/consent/assent (e.g., terminally ill receiving hospice services, and/or receiving post-hospital skilled rehabilitation) that may not allow enough time for obtaining consent/assent, and scheduling days for video recording sessions across three-time points (baseline, and 6- and 12- weeks post-baseline)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liu Wen, PhD, Principal Investigator — The University Of Iowa College Of Nursing
Locations (1):
- Iowa Vateran's Home, Marshalltown, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Families were to be recruited for Aim 1 only to collect feedback on OPTIMAL. We recruited 94 staff, much more than we planned (20 staff) and were able to collect adequate feedback from 94 staff on OPTIMAL for refinement. Our team agreed to move to Aim 2 and 3 (testing OPTIMAL in NH staff and residents) and we did not enroll families as participants but engaged some families of resident participants as community stakeholders (vs. participants/subjects) in refining OPTIMAL.
Pre-assignment Details: A total of 111 participants (94 staff, 17 residents) were enrolled at baseline, 1 resident lost to follow up at data collection time point 2, resulting in a total of 110 participants who retained in follow up data collections.
Groups:
- Residents: Resident participants who were cared in the study site, and received care from the staff participants before and after the OPTIMAL intervention was delivered to staff.
Period: Overall Study
Arm/Group | Staff | Residents
Started | 94 | 17
Completed | 94 | 16
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm1: OPTIMAL
  OPTIMAL: A person-centered mealtime care intervention.
Arm/Group | Arm1
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 111 participants (overall number) = 17 resident participants + 94 staff participants
  years
    Resident participants: number analyzed (Participants) | 17
    Resident participants | 73.9 (7.9)
    Staff Participants: number analyzed (Participants) | 94
    Staff Participants | 44.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 111 participants (overall number) = 17 resident participants + 94 staff participants
  Participants
    Resident participants: number analyzed (Participants) | 17
    Resident participants: Female | 2
    Resident participants: Male | 15
    Staff participants: number analyzed (Participants) | 94
    Staff participants: Female | 86
    Staff participants: Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 111 participants (overall number) = 17 resident participants + 94 staff participants
  Participants
    resident participants: number analyzed (Participants) | 17
    resident participants: While | 15
    resident participants: Non white | 2
    staff participants: number analyzed (Participants) | 94
    staff participants: While | 82
    staff participants: Non white | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 111
Education Level [Count of Participants; unit: Participants] — Population: 111 participants (overall number) = 17 resident participants + 94 staff participants
  Participants
    Resident Participants: number analyzed (Participants) | 17
    Resident Participants: up to high school | 3
    Resident Participants: some college/college graduate/post-college | 4
    Resident Participants: don't know/refused | 10
    Staff Participants: number analyzed (Participants) | 94
    Staff Participants: up to high school | 32
    Staff Participants: some college/college graduate/post-college | 37
    Staff Participants: don't know/refused | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Staff Participants Who Viewed the Intervention as Appropriate and Acceptable for Mealtime Care Practice
Description: All staff participants were interviewed on whether the intervention protocol and training materials were acceptable and appropriate for nursing home mealtime care practice before pilot testing.
Time Frame: After recruitment of staff participants and before T1 (baseline)
Population: Only the staff arm/group was assessed for this outcome measure, because only staff participants received training materials and training sessions directly from research team. In addition, the "residents" arm/group consisted of people living with moderate-to-severe dementia and were not able to provide accurate and valid information regarding whether the intervention protocol and training materials were acceptable and appropriate for nursing home mealtime care practice.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff
Number analyzed (Participants) | 94
Participants | 94

2. Primary Outcome: Number of Staff and Resident Participants Recruited and Retained for the Study
Description: The number of staff and resident participants that were recruited at baseline and retained over the study period were collected to indicate the feasibility of the study on participant recruitment, consent and retention.
Time Frame: From recruitment/consent throughout the study completion, up to 12-weeks post baseline
Population: These are the number of staff and resident participants that were recruited at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Staff | Residents
Number analyzed (Participants) | 94 | 17
Participants | 94 | 16

3. Primary Outcome: The Number of Staff Participants Who Attended All Training Sessions
Description: A checklist was used to track the number of staff participants who attended all the group and/or individual training sessions that were provided in the study.
Time Frame: During each OPTIMAL training session (within 2 weeks post baseline)
Population: All 94 staff participants attended all the training sessions provided during the study
Measure: Count of Participants; unit: Participants
Arm/Group | Staff
Number analyzed (Participants) | 94
Participants | 94

4. Primary Outcome: Staff Person-centered Care Knowledge and Self-efficacy
Description: Training receipt, indicated by a total score of ≥ 75% on the staff PCMC-related knowledge & self-efficacy test post-training with or without booster sessions. The total score of the scale ranges from 0 - 20, and higher scores are better. we recorded the number of staff who reached this cutoff score post training.
Time Frame: Right before and after OPTIMAL training session (within 2 weeks post baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Staff
Number analyzed (Participants) | 94
Participants | 94

5. Primary Outcome: Number of Staff Participants Who Viewed the Intervention Was Useful
Description: All staff participants were interviewed on whether the intervention was useful post testing. The number of staff participants who viewed the intervention was useful was collected.
Time Frame: After T3 data collection time point (12-weeks post baseline)
Population: All 94 staff participants were interviewed on whether the intervention was useful post testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff
Number analyzed (Participants) | 94
Participants | 94

6. Primary Outcome: The Number of Mealtime Difficulty Behaviors Observed in Residents
Description: Videos will be coded using the Cue Utilization and Engagement in Dementia (CUED) mealtime video coding scheme that have codes for resident mealtime difficulties including 1) resistive behaviors and 2) functional impairments. we recorded the number of behaviors representing mealtime difficulties presented by residents, the higher the number, the worse the outcome.
Time Frame: T1 (baseline), T2 (6-weeks post baseline), T3 (12-weeks post baseline)
Measure: Mean (Standard Deviation); unit: number of mealtime difficulty behaviors
Arm/Group | Residents
Number analyzed (Participants) | 16
number of mealtime difficulty behaviors
  Baseline | 6.5 (4.6)
  Week 6 | 2.5 (2.9)
  Week 12 | 4.2 (2.8)

7. Primary Outcome: Resident Level of Eating Performance
Description: Level of Eating Independence Scale, a 9-item scale assessing the ability of independence with eating and drinking activities during cycles of verbal prompts, will be used to measure. Each item is scored from 1 (total dependence) to 4 (total independence), with total score ranging from 9 to 36 (higher score = more independence).
Time Frame: T1 (baseline), T2 (6-weeks post baseline), T3 (12-weeks post baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Residents
Number analyzed (Participants) | 16
score on a scale
  Baseline | 31 (6)
  Week 6 | 28.4 (8.4)
  week 12 | 27.4 (8.8)

8. Primary Outcome: Resident Intake Success Rate
Description: Videos will be coded using CUED to track whether the resident or staff initiates/completes each intake attempt and whether there is a subsequent intake after each attempt. Resident intake success rate will be calculated by dividing the number of intake attempts initiated/completed by the resident with subsequent intake by the total number of intake attempts coded during one meal. the percent can range from 0 - 100%, the higher the number, the more independent the resident.
Time Frame: T1 (baseline), T2 (6-weeks post baseline), T3 (12-weeks post baseline)
Measure: Mean (Standard Deviation); unit: percentage of resident successful intake
Arm/Group | Residents
Number analyzed (Participants) | 16
percentage of resident successful intake
  Baseline | 94.3 (7.3)
  Week 6 | 92.2 (7.7)
  Week 12 | 91.1 (9.7)

9. Secondary Outcome: Quality of Staff Engagement
Description: Quality of staff engagement will be assessed by Mealtime Engagement Scale developed by the PI with evidence of reliability and validity (each item is scored on 0-3, total score range: 0-57, higher score = higher quality of engagement).
Time Frame: T1 (baseline), T2 (6-weeks post baseline), T3 (12-weeks post baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff
Number analyzed (Participants) | 94
score on a scale
  Baseline | 24.2 (14.4)
  Week 6 | 13.9 (6.3)
  Week 12 | 16.3 (5.9)

10. Secondary Outcome: Resident Body Mass Index (BMI).
Description: Resident Body Mass Index (BMI, unit is kg/m2). We will assess body weight in the early morning before breakfast with each individual resident dressing casual indoor clothes without shoes using the same digital body scale throughout the study. We will assess body weight twice in one early morning of each time point and calculate the average of the two assessments for BMI.
Time Frame: T1 (baseline), T2 (6-weeks post baseline), T3 (12-weeks post baseline)
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Residents
Number analyzed (Participants) | 16
kg/m2
  Baseline | 30.9 (5.1)
  Week 6 | 30.1 (5.3)
  Week 12 | 30.1 (5.9)

ADVERSE EVENTS:
Time Frame: Adverse event were collected at 3 time points: baseline (T1), immediately post intervention (6 weeks post baseline, T2), and 6-week post intervention (12 weeks post baseline, T3).
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, is not different from the clinicaltrials.gov Definitions.
Groups:
- Families: In this study, we were initially planning to recruit families for our Aim 1 to collect feedback on the OPTIMAL intervention. The fact that we recruited 94 staff (initially planned for 20 staff recruitment), which is much more than we planned, and we were able to collect feedback from these staff on the OPTIMAL intervention which helped refinement of the intervention. Our team agreed that we received adequate feedback to move to Aim 2 and 3 (testing the OPTIMAL intervention in NH staff and residents, where families were not included in the proposed study). Therefore, we did not enroll families as participants, but communicated with them regarding the refined OPTIMAL and engaged N=5 family members in this effort where they served as community stakeholders and no individual characteristics were needed to be collected (rather than study participants/subjects who need to consent to be enrolled and followed up over time).
Arm/Group | Staff | Residents | Families
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/17 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/17 | 0/0
Other Adverse Events (participants affected / at risk) | 0/94 | 0/17 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT05255068/Prot_SAP_000.pdf